CLINICAL TRIAL: NCT05255432
Title: Summative Evaluation to Validate That the Laryngeal, Endo-tracheal, Airway Fixator (LEAFix) Can be Used Safely and Effectively by Intended Users to Secure Airway Devices
Brief Title: Summative Evaluation to Validate the LEAFix Device With Users
Acronym: LEAFIXUser
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: SP0920
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Selection of tasks
  Interventions: Other: nil intervention
- Group B: Selection of tasks
  Interventions: Other: nil intervention

INTERVENTIONS:
Other: nil intervention — Users observation using medical device on manakin, different scenarios per group

SUMMARY:
The Laryngeal Endo-tracheal Airway Fixator(LEAFix) is a single use product designed to secure airway devices to patients during anaesthesia, with better infection control management and interaction with the patients skin. This study investigates the users of the LEAFix device interacting with the LEAFix device, its packaging and a simulated patient through different scenarios of securing an airway device. The aim is to understand the risks associated with the use of the device for CE marking purposes. This study is funded by Innovel Ltd. the manufacturer of the device.

ELIGIBILITY:
Inclusion Criteria:

* Member of staff trained in placing airways

Exclusion Criteria:

* Previous knowledge of the device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practioners who perform airway placement
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Performance of user against the predetermined standard | 1 hour
  The users will be marked against a standard set to look for problems

IPD SHARING:
Plan to Share IPD: No